CLINICAL TRIAL: NCT04165148
Title: Randomized Study Comparing the Low Impact Laparoscopy Concept to Conventional Laparoscopy in Terms of Ambulatory Care
Brief Title: Low Impact Laparoscopy Concept Versus Conventional Laparoscopy
Acronym: RANDOLIL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no more material
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0335; 2019-A01863-54 (Other: ID-RCB)
Record Dates: First submitted 2019-11-07; First posted 2019-11-15 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Ambulatory Laparoscopic Hysterectomy
Keywords: Low Impact Laparoscopy; laparoscopy; hysterectomy; ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Impact Laparoscopy (Experimental): Low Impact Laparoscopy is a minimally invasive technique that combines low pressure insufflation (with the Intelligent Flow System (iFS) AirSeal® system) and microcoelioscopy (with specific microtrocards and laparoscopic instruments).
  Interventions: Device: Low Impact Laparoscopy; Other: Visual Analog Scale (VAS) for Pain; Other: Saint-Antoine Pain Questionnaire (QDSA); Other: post-operative questionnaire
- conventional laparoscopy (Active Comparator): conventional laparoscopy
  Interventions: Device: conventional laparoscopy; Other: Visual Analog Scale (VAS) for Pain; Other: Saint-Antoine Pain Questionnaire (QDSA); Other: post-operative questionnaire

INTERVENTIONS:
Device: Low Impact Laparoscopy — Low Impact Laparoscopy is a minimally invasive technique that combines low pressure insufflation (with the iFS AirSeal® system) and microcoelioscopy (with specific microtrocards and laparoscopic instruments).
  Arms: Low Impact Laparoscopy
Device: conventional laparoscopy — conventional laparoscopy
  Arms: conventional laparoscopy
Other: Visual Analog Scale (VAS) for Pain — The patient evaluates her pain using an VAS scale on arrival in the post-interventional surveillance room, then 30 minutes, 2 hours, 4 hours, 6 hours after leaving the operating roo, at the exit of post-interventional surveillance room and at the exit of the hospital.
  The day after surgery, according to the usual practice, outpatients receive a telephone call from a Gynecologist. The assessment of their pain (with VAS scale) will be collected.
  During the usual consultation at 1 month, the patient must evaluate her pain by means of an VAS.
Other: Saint-Antoine Pain Questionnaire (QDSA) — The patient evaluates her pain using an QDSA questionnaire on arrival in the post-interventional surveillance room, then 30 minutes, 2 hours, 4 hours, 6 hours after leaving the operating roo, at the exit of post-interventional surveillance room and at the exit of the hospital.
  The day after surgery, according to the usual practice, outpatients receive a telephone call from a Gynecologist. The assessment of their pain (with QDSA questionnaire) will be collected.
  During the usual consultation at 1 month, the patient must evaluate her pain by means of an QDSA questionnaire.
Other: post-operative questionnaire — The patient will fill in the antalgic intake record and the patient booklet for the collection of medical consumptions from her discharge from the hospital and during the month following the surgery.

SUMMARY:
Outpatient surgical management has been developing in recent years and High Authority of Health recommendations in French for this type of management is a postoperative pain score of less than 3 on the VAS.

The feasibility and safety of laparoscopy is well established, particularly in the field of gynecology, but this technique often causes postoperative pain. Techniques are being developed to reduce postoperative pain in laparoscopic surgery. Low pressure insufflation (7 to 10 mmHg) compared to standard pressure insufflation (12 to 15 mmHg) significantly reduces postoperative pain. Microcoelioscopy (use of 3 mm trocars instead of 5 to 12 mm trocars in standard laparoscopy), by reducing the size of incisions, also significantly reduces postoperative pain.

The Low Impact Laparoscopy is a minimally invasive technique that combines low pressure insufflation and microcoelioscopy which would have the advantage of reducing postoperative pain. This technique would therefore, by reducing postoperative pain, to improve outpatient management, particularly in cases of hysterectomies for which the outpatient management rate could be increased.

The hypothesis is that using the Low Impact Laparoscopy concept would increase outpatient management rate compared to conventional laparoscopy in gynecological surgeries for hysterectomy.

The study aims to compare the Low Impact Laparoscopy concept with conventional laparoscopy in terms of ambulatory care rates in patients undergoing surgery for hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years
* planned surgery procedure : ambulatory laparoscopic hysterectomy
* effective contraception if women of childbearing age
* patients with free, informed and signed consent

Exclusion Criteria:

* disorders leading to an unacceptable risk of postoperative complications sought during the interrogation of the patient (disorders of blood coagulation, disorders of the immune system, progressive diseases ....)
* pregnancy or wish for subsequent pregnancy
* lactating women
* contraindication to laparoscopy
* contraindication to minimally invasive endoscopic techniques
* not eligible for outpatient care
* inability to understand the information given
* a person not affiliated to a social security scheme, or deprived of liberty, or under guardianship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
success rate of ambulatory care | 1 month after surgery
  rate of patients actually managed on an outpatient setting (discharged from hospital the same day of the intervention) and who presented no complication or rehospitalization in the month following the intervention

SECONDARY OUTCOMES:
pain score (Visual analogic scale (VAS) for pain) | arrival in the post-interventional surveillance room
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | 30 minutes after exit of operating room
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | 2 hours after exit of operating room
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | 4 hours after exit of operating room
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | 6 hours after exit of operating room
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | at the exit of a post-interventional surveillance room, an average of 2 hours after arrival
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | on leaving the hospital, an average of 8 hours after surgery
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | the day after surgery
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (VAS) | 1 month after surgery
  Visual analogic scale (VAS) is used to evaluate from 0 (no pain) to 10 (unbearable pain)
pain score (Saint-Antoine Pain Questionnaire (QDSA questionnaire)) | 6 hours after exit of operating room
  Pain score assessed by QDSA short questionnaire (Saint-Antoine Pain Questionnaire) : list of 16 qualifiers to describe pain, score ranging from 0 to 64.
pain score (Saint-Antoine Pain Questionnaire (QDSA)) | the day after surgery
  Pain score assessed by QDSA short questionnaire (Saint-Antoine Pain Questionnaire) : list of 16 qualifiers to describe pain, score ranging from 0 to 64
dose of morphine | at the exit of a post-interventional surveillance room, an average of 2 hours after arrival
  total dose of morphine (miligramme (mg)) administered in the post-interventional surveillance room
number of patients who needed an analgesic | at the exit of a post-interventional surveillance room, an average of 2 hours after arrival
  number of patients who needed an analgesic supplement in post-interventional monitoring room
number of patients who needed an analgesic | on leaving the hospital, an average of 8 hours after surgery
  number of patients who needed an analgesic supplement in post-interventional monitoring room
number of patients who needed an analgesic | 1 month after surgery
  number of patients who needed an analgesic supplement in post-interventional monitoring room
total administered dose | at the exit of a post-interventional surveillance room, an average of 2 hours after arrival
  total administered dose of analgesic supplement (mg) in post-interventional monitoring room
total administered dose | on leaving the hospital, an average of 8 hours after surgery
  total administered dose of analgesic supplement (mg) in post-interventional monitoring room
total administered dose | 1 month after surgery
  total administered dose of analgesic supplement (mg) in post-interventional monitoring room
duration of analgesic treatment | on leaving the hospital
  duration of analgesic treatment (days) during the hospital stay
duration of analgesic treatment | 1 month after surgery
  duration of analgesic treatment (days) during the hospital stay
operating time | at the exit of the operating room, an average of 30 minutes after surgery
  operative time (between incision and closure) in minutes
number of per and postoperative complications | 1 month after surgery
  number of per and postoperative complications
types of per and postoperative complications | 1 month after surgery
  description of per and postoperative complications
hours total of stay in the post-intervention monitoring room | at the exit of a post-interventional surveillance room
  length of stay in the post-interventional surveillance room in hours
number of days of hospital stay | on leaving the hospital
  length of hospital stay (if non ambulatory care) in number of days
number of days of work stoppage | 1 month after surgery
  duration of work stoppage of the patient in number of days
patient management costs | 1 month after surgery
  Patient management costs according to the two surgical strategies

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France